Official title: Effect of Low Carbohydrate Versus Low Fat Diet in the Treatment of Dyslipidemia

in Obese Children with Metabolic Syndrome

NCT number: NCT03937960 Document date: 10/06/2022

Primary grant number: NIH P30 - DK056336

Sample Size: Selected per budgetary constraints for a pilot grant.

Student's t-test and Mann-Whitney test will be used to compare variables for continuous parametric and non-parametric variables respectively. The chi-square test will be used to compare categorical variables. Spearman correlations (r) will be used to compare continuous variables. Bivariate correlations will be calculated between vascular outcome variables and lipid parameters overall and by group. Exploratory general linear models will be used to explore lipid and lipoprotein profile assays. We will plan to adjust for covariates: age, sex, insulin treatment, duration of diabetes and glycemic control if possible. P<0.05 will be considered statistically significant.